CLINICAL TRIAL: NCT01059747
Title: Therapeutic Drug Monitoring and Pharmacogenomics Study of Methadone Therapy
Acronym: M0108
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Keh-Ming Lin, Director, Division of Mental Health and Addiction Medicine, National Health Research Instiutes, Taiwan
Other Study IDs: 98A1-PHPP41
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Last update posted 2010-02-01 (Estimated); Status verified 2010-01

CONDITIONS: Heroin-addicted Patients Who Undertook Methadone Maintenance Treatment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- treatment group
  Interventions: Other: no intervention applied

INTERVENTIONS:
Other: no intervention applied — no intervention applied

SUMMARY:
Addiction has been regarded as one of the most serious health and social problems in Taiwan, and heroin is currently considered to be the major substance of abuse. The most widely used treatment to date is methadone replacement therapy. It is reported that to achieve a better clinical response and to avoid possible side effects, the blood level of methadone should remain in a certain level. However, the blood level of methadone is mediated by various factors besides dosage. Genetic variability in genes that encodes enzymes affecting methadone metabolism, target receptors of methadone, and drug-drug interaction by other medication patients take will all affect blood level. Therefore, therapeutic drug monitoring (TDM) and pharmacogenomic study is crucial for evaluating and predicting the clinical response, cause of side effects or toxicity, as well as studies on drug-drug interactions.

This is a cross-sectional study in order to evaluate the relationship between methadone plasma level and clinical response in patients under methadone maintenance therapy and to identify optimal therapeutic thresholds. HPLC will be used to analyze methadone and its metabolites. Our hypothesis is that methadone plasma levels in patients who are responsive to methadone maintenance therapy are higher than level in non-responsive patients, and higher plasma level leads to less severe withdrawal symptoms. We will also test if an optimal minimal dosage exists among these patients. In the meanwhile, we will aim to test if methadone level and clinical response is correlated with different genetic polymorphism. Candidate genes that involve in pharmacokinetic and pharmacodynamic process of methadone (e.g. CYP3A4, CYP3A5, CYP2B6, ABCB1, opioid mu receptor and kappa receptor) will be genotyped for these analyses.

The results of this study will provide clinical information of methadone treatment and pharmacogenomic data in Taiwanese for clinicians to achieve a better treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese ethnicity
2. Men or women above age of 18
3. Able to participate in a clinical assessment in Chinese (including Mandarin and Taiwanese dialects)
4. Diagnosis of Heroin dependence by DSM-IV definition
5. Enter methadone maintenance therapy for at least 3 months
6. No change of methadone dosage for the last week
7. Regularly took methadone for the last week
8. Individuals who have completed a written consent form

Exclusion Criteria:

1. Patients with comorbid severe mental disorders including:

   1. Organic mental disorders, or
   2. Schizophrenia
2. Severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: heroin-addicted patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Chang Wang, MD, Principal Investigator — National Health Research Institutes, Taiwan
Locations (7):
- Taiwan (7):
  - Departments of Psychiatry, Wei-Gong Memorial Hospital, Miaoli
  - Departments of Psychiatry, China Medical University and Hospital, Taichung
  - Departments of Psychiatry, Taipei City Hospital Song-De Campus, Taipei
  - Departments of Psychiatry, Taipei City Hospital Yang-Ming Campus, Taipei
  - Departments of Psychiatry, En-Chu-Kong Hospital, Taipei County
  - Departments of Psychiatry, Far-Eastern Memorial Hospital, Taipei County
  - Departments of Psychiatry, Tao-yuan Psychiatric Center, Taoyuan District

REFERENCES:
- [Derived] Liu SW, Liu YL, Hwang LL, Wang SC, Kuo HW, Wu SL, Dai YW, Liu SC, Ho IK, Chen AC, Hsiao CF, Tsou HH. Chemokine IP-10 is correlated with cardiac responses and status of infection with HIV and HCV in methadone maintenance patients. Int J Cardiol. 2015 Sep 1;194:36-8. doi: 10.1016/j.ijcard.2015.05.055. Epub 2015 May 12. No abstract available. PMID 26011262
- [Derived] Tsai HJ, Wang SC, Tian JN, Chang TK, Ho IK, Hsiao CF, Chen CH, Tan HK, Lin L, Wu CS, Su LW, Huang CL, Yang YH, Liu ML, Lin KM, Liu YL. PXR polymorphisms interacted with CYP2B6 polymorphisms on methadone metabolites. J Clin Psychopharmacol. 2013 Feb;33(1):137-40. doi: 10.1097/01.jcp.0000426186.34421.de. No abstract available. PMID 23288240
- [Derived] Wang SC, Tsou HH, Chen CH, Chen YT, Ho IK, Hsiao CF, Chou SY, Lin YF, Fang KC, Huang CL, Su LW, Fang YC, Liu ML, Wu HY, Lin KM, Liu SC, Kuo HW, Chiang IC, Chen AC, Tian JN, Liu YL. Genetic polymorphisms in the opioid receptor mu1 gene are associated with changes in libido and insomnia in methadone maintenance patients. Eur Neuropsychopharmacol. 2012 Oct;22(10):695-703. doi: 10.1016/j.euroneuro.2012.02.002. Epub 2012 Mar 9. PMID 22406240